CLINICAL TRIAL: NCT06186011
Title: Quality of Life and Cosmetic Outcomes of Breast-Conserving Surgery According to Localization Method (TRIGUIDE Trial) - A Randomized Trial
Brief Title: Quality of Life and Cosmetic Outcomes of Breast-Conserving Surgery According to Localization Method
Acronym: TRIGUIDE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCB/2023/0141
Record Dates: First submitted 2023-12-15; First posted 2023-12-29 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-10

CONDITIONS: Breast Cancer
Keywords: Quality of Life; Cosmetic outcomes
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Single-center parallel randomized Clinical Trial with three arms: intraoperative Ultrasound vs. wire vs. radioactive seed
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Wire-guided (Active Comparator): Wire guided localization (WGL) is considered the standard method for intraoperative localization of non-palpable breast lesions, chosen by many centers worldwide. It involves the placement of a wire or barbed needle that is percutaneously introduced into the lesion using a guide. It is cost-effective, easy to place guided by ultrasound or stereotaxis, allows for repositioning in case of error, and its safety and efficacy have been widely demonstrated in the literature.
  Interventions: Procedure: Wire-guided surgery
- Intraoperative Ultrasound (Active Comparator): The use of intraoperative ultrasound (IOUS) is an effective method that is controlled by the surgeon and does not require the involvement of other departments or preoperative invasive procedures. IOUS has been introduced into clinical practice as a tool for visualizing non-palpable tumors, demonstrating the detection of nearly 100% of lesions, and a rate of negative margins and re-excision similar to WGL. One of the challenges of the technique in ultrasound-guided surgery arises when the tumor is <5mm, making it difficult to visualize by ultrasound, or when there are microcalcifications not visible by ultrasound.
  Interventions: Procedure: Intraoperative ultrasound localization
- Radioactive seed (Active Comparator): Radioactive seeds are composed of a titanium capsule with an I-125 filament inside. They have low radioactivity, which can range from 7 to 200 μCi. During surgery, the seeds are detected using a portable gamma ray detection probe typically used for sentinel lymph node biopsy, configured to detect an I-125 source (27 keV). This probe has a wide detection range through tissue (>10 cm), currently offering the greatest detection range compared to other available localization devices. Radioactive seed localization (RSL) require coordination between the radiology and nuclear medicine departments for marking. The results in terms of lesion localization and margin involvement rates are comparable to WGL.
  Interventions: Procedure: Radioactive seed localization

INTERVENTIONS:
Procedure: Wire-guided surgery — If assigned to the WGS, the marking will be performed by the radiologist on the day prior to the intervention.
  Arms: Wire-guided
Procedure: Radioactive seed localization — If assigned to the RSL, the marking will be performed by the radiologist on the day prior to the intervention. The handling and traceability will be done by the nuclear medicine physician.
  Arms: Radioactive seed
Procedure: Intraoperative ultrasound localization — If the patient is assigned to the Intraoperative ultrasound localization (IOUS), no further procedures will be necessary until surgery. Subsenquently, the primary surgery will be performed.
  Arms: Intraoperative Ultrasound

SUMMARY:
The goal of this clinical trial is to compare Quality of Life and cosmetic outcomes in Breast Conservative Carcer surgery depending on localization method (intraoperative Ultrasound, wire and radioactive seed).

Participants will be randomly assigned to one of the three proposed arms, and the primary surgery will be performed.

DETAILED DESCRIPTION:
INTRODUCTION:

The surgery for breast cancer is increasingly emphasizing cosmetic outcomes, body image, and the quality of life (QoL) of patients. Survival is the top priority; however, other concerns or problem areas may arise, such as dissatisfaction with body image. All of this has implications for QoL, self-esteem, relationships, and sexual functionality. One of the challenges of breast conservative surgery (BCS) is suboptimal cosmetic results, which can be observed in up to 40% of patients in some series. Factors influencing the cosmetic outcome include patient characteristics such as weight or breast density, the volume of the tumor removed, the tumor's location in the breast, wound complications, and the dose and schedule of radiotherapy. Therefore, the use of low-visibility incisions, precise tumor resection, and the introduction of oncoplastic techniques have revolutionized the surgical management of these patients.

The localization of the lesion is a key point for surgical resection. Advancements in imaging diagnostic methods and molecular classification have led to a reevaluation of surgical approaches. The widespread use of mammography as a screening method for breast cancer has resulted in an increase in the detection of non-palpable breast lesions, necessitating the search for tools to detect these lesions. The intent of surgery should always be both radical and effective, meaning achieving the removal of the loco-regional disease. The main challenge in breast surgery lies in striking a balance between wide excision with clear margins and a satisfactory cosmetic outcome Currently, there are multiple localization techniques available, although the evidence from comparative studies is limited. Wire guided localization (WGL) is considered the standard method for intraoperative localization of non-palpable breast lesions and is the method of choice for many centers worldwide. However, alternative localization techniques such as radioguided occult lesion localization using radioactive iodine-125 seeds (RSL) and ultrasound guided surgery (UGS) have recently been shown to reduced re-excision rates. In a systematic review comparing different localization methods, UGS reduced the percentage of involved margins and significantly decreased the reoperation rate and surgical time when compared to WGL. UGS also showed a statistically significant reduction in the number of involved margins compared to RSL. All techniques were equivalent in terms of effectiveness, localization complications, and general complications. The available evidence on cosmetic outcomes and QoL in BCS according to the localization technique is limited.

We hypothesized UGS and RSL would be associated with a better QoL and cosmetic outcome compared to WGL. The aim of TRIGUIDE study was to compare the QoL and cosmetic outcomes of women who underwent BCS according the localization method.

METHOD/PROCEDURES:

All eligible patients scheduled for primary surgery with ecovisible lesions will be prospectively recruited from external Gynecology consultations. They will have attended the consultation according to the usual care pathway, after completing complementary tests and receiving a confirmed diagnosis. An ultrasound will be performed by the surgeon in the consultation to confirm the identification of the lesion. Baseline quality of life (QoL) will be assessed using the BREAST-Q questionnaire (preoperative).

The surgical procedure will be jointly decided by the surgeon and the patient and will not be modified by the study. Patients will be consecutively and randomly assigned to one of the three proposed arms. If the patient is assigned to the intraoperative ultrasound arm, no further procedures will be necessary until the surgery. If assigned to the wire or seed arm, the marking will be performed by the radiologist on the day prior to the intervention. The handling and traceability of the radioactive seed, if applicable, will be done by the nuclear medicine physician. Subsequently, the primary surgery will be performed. We will preserve the orientation of the specimen with marking sutures, such that positive resection margins could be identified and re-excised if necessary. Radiological margin assessment will be conducted during procedure and ampliations will be performed with the advice of the radiologist and the surgeon's discretion. We will undertake axillary surgery in the same session, according to international guideline. The surgical specimen will be postoperative processed and analyzed by the Pathology Department. A multi- disciplinary team will review all cases preoperatively and postoperatively, and we will administer adjuvant radio- therapy or systemic therapy according to institutional and national guidelines. Regular follow-up will be carried out by the Gynecology team, with a visit at 3-4 weeks and 12 months post-surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with non-palpable and ecovisible infiltrating breast carcinoma, classified as T1 and T2, eligible for primary breast-conserving surgery (BCS)

Exclusion Criteria:

* lesions <5mm
* multicentric tumors
* extensive calcifications not visible by ultrasound
* level III oncoplastic techniques or mastectomy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-10-04 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
BCCT.core | 12 months after surgery
  BCCT.core is a semi-automatic software validated for the assessment of cosmetic outcomes following BCS. It provides an objective measure and has been demonstrated to correlate well to a panel of experts. BCCT.core analyses several parameters including symmetry, skin colour and scar visibility to evaluate breast cosmesis, and classifies the overall cosmetic result into four classes: Excellent, Good, Fair and Poor. However, BCCT.core does not incorporate patient self-perception of outcome and does not directly assess the volume of breast excised. Standardized clinical photographs were taken 1-year post-surgery with or without radiotherapy, as recommended by the BCCT.core software developers and assessed at the end of the data collection period by a single investigator, blinded to the identification and treatment group of the participant.
BREAST-Q questionnaire | preoperative, 12 months after surgery
  The BREAST-Q questionnaire is a specific and validated Patient-Reported Outcome Measure (PROM) for patients undergoing breast surgery designed to assess the outcomes and satisfaction of individuals, which measures health-related QoL (physical well-being, psychological and sexual) and satisfaction (satisfaction with the breast, satisfaction with the overall result and satisfaction with the care received). Each scale is scored to generate a numeric score on a scale from 0 (worst) to 100 (best). These measures were studied at baseline (preoperative) and 12 months post-surgery.

SECONDARY OUTCOMES:
Excess volume resection | Inmediatly after surgery
  Defined by the resected breast volume minus the tumor volume
Margin status | Inmediatly after surgery
  negative - no tumour cells at inked margin; or positive - tumour at the inked edge
Ampliations | Inmediatly after surgery
  Number of ampliations to reach negative margin status
Additional treatment interventions | 3 weeks and 12 months after surgery
  Record the need for new surgeries, both for margin ampliation and complications
Excision time | Inmediatly after surgery
  defined in min as the time from the first mammary incision to wound closure
Postoperative complications | Inmediatly after surgery, 3 weeks and 12 months after surgery
  Seroma, hematoma, infection and their management (conservative, drainage, antibiotic therapy, drainage)
Surgeon satisfaction | Inmediatly after surgery
  Surgeon satisfaction with localization method with a Likert scale:
  1. - Very dissatisfied
  2. - Dissatisfied
  3. - Unsure
  4. - Satisfied
  5. - Very satisfied

CONTACTS AND LOCATIONS:
Overall Officials: Eduard Mension, MD PhD, Principal Investigator — Hospital Clinic of Barcelona
Locations (1):
- Hospital Clínic de Barcelona, Barcelona, Spain